CLINICAL TRIAL: NCT00462618
Title: Group Cognitive Behavioral Therapy (CBT I) Vs. Quetiapine for Residual Insomnia Impairing Recovery Among Elderly With Stable Major Affective Disorders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rayan Al Jurdi, MD, PI, Michael E. DeBakey VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-19343
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Insomnia
Keywords: Insomnia; Elderly; Affective disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Mood Disorders | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBT (Active Comparator)
  Interventions: Drug: Quetiapine; Behavioral: Cogntive behavioral therapy

INTERVENTIONS:
Drug: Quetiapine
Behavioral: Cogntive behavioral therapy

SUMMARY:
The purpose of this pilot study is to assess feasibility and patient accessibility in order to design an adequately powered study to compare group cognitive behavioral therapy for insomnia (CBT-I) to quetiapine in non-demented patients aged 60 years or older with controlled bipolar disorder (I or II) or major depressive disorder who suffer from residual insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater or equal to 60 years.
2. Patients with history of major affective disorder, including Bipolar disorder type I or type II or major depressive disorder, as assessed by the Structured Clinical Interview for DSM-IV (SCID), currently in remission.
3. Difficulty starting or initiating sleep four or more times/week for at least 3 months by history.
4. Total Pittsburg Sleep Quality Index >5.

Exclusion Criteria:

1. Patient in an acute mood episode as assessed by SCID
2. Patients with sleep disruptive medical problems including: sleep apnea, restless leg syndrome, periodic limb movement, parasomnia, congestive heart failure, chronic pain and chronic obstructive pulmonary disease as assessed by medical history and medical record review.
3. Patients with schizophrenia, primary anxiety disorder and active substance abuse as determined by SCID.
4. Patients on or with history of failure or intolerance to respond to quetiapine.
5. Patient with positive Alcohol Use Disorders Identification Test (AUDIT) with a total score above 8.
6. Patients with dementia brain degenerative diseases, cognitive disorders and Mini Mental Status Examination (MMSE) score of less or equal to 24.
7. Patients who are in an acute depressive, manic, hypomanic or mixed state as reflected by SCID
8. Patients on concurrent sedating medications that would confound interpretation of the results. This is operationalized as follow: Sedating medications must be present and stable dosage for at least 14 days prior to enrollment in the study. If the medication is not prescribed as a primary sleep aid, it will be continued. Our rationale is that patients may need these medications and the initial sedating effect will have plateaued by 14 days. However, medications prescribed to assist insomnia will be discontinued as they are not effective for the subjects who otherwise meet inclusion ad exclusion criteria for the current study. Medications will be tapered as clinically indicated after the patients sing informed consent and prior to baseline assessment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
PTSQ | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rayan k Al Jurdi, Principal Investigator — Michael Debakey VAMC, Baylor College of Medicine
Locations (1):
- Michael Debakey VAMC, Houston, Texas, United States